CLINICAL TRIAL: NCT03792360
Title: A Pilot Study: Evaluating the Safety and Feasibility of Using Autologous Adipose-Derived Stromal Vascular Fraction (SVF) for the Treatment of Aerodigestive & Enterocutaneous Fistulae in Adults
Brief Title: Adipose Derived SVF for Aero-digestive & Enterocutaneous Fistulae
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed due to lack of patient enrollment.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Bhaumik Brahmbhatt, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-003774
Record Dates: First submitted 2018-11-21; First posted 2019-01-03 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Tracheoesopharyngeal Fistula; Bronchoesophageal Fistula; Tracheoesophageal Fistula
MeSH Terms: conditions — Tracheoesophageal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: SVF (Stromal Vascular Fraction)

INTERVENTIONS:
Drug: SVF (Stromal Vascular Fraction) — The stromal vascular fraction (SVF), isolated when fresh lipoaspirates are enzymatically digested with a collagenase, contains a heterogeneous cellular and extracellular milieu. SVF is an aqueous fraction, consisting of endothelial cells and their precursors, macrophages, smooth muscle cells, lymphocytes, pericytes, pre-adipocytes and actual AMSCs.

SUMMARY:
Determine safety and feasibility of using institutionally prepared autologous, uncultured SVF on patients with aerodigestive and enterocutaneous fistulae secondary to malignancy, trauma or surgery.

DETAILED DESCRIPTION:
The primary aim of this pilot study is to evaluate the feasibility, time, cost, safety, limitations, and efficacy of the use of institutionally processed SVF for management and closure of aero-digestive and enterocutaneous fistulae. This pilot study would help identify design issues and the potential success of fistulae closure by the means of autologous SVF administration before a full-scale trial is performed.

A secondary aim is the closure of aero-digestive and enterocutaneous fistulae along with characteristics such as size, etiology, recurrence, localization, and the association of these factors withoutcome after SVF administration. The SVF quantification, characterization and differentiation in vitro will be described.

This process will help identify the type of fistulae that are susceptible to closure with human cell therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years old
* Adults ≤ 90 years old
* Fistula or sinus tract opening size between 2 mm and 15 mm in diameter (as measured by comparing its size with the open mouth of a biopsy forceps)
* Inpatient or outpatient setting
* Recurrent or de novo fistulas or sinus tracts
* A prior diagnosis of ADF OR ECF in which the standard therapy has failed or is not applicable
* Fistula or sinus tract location may include:
* Tracheopharyngeal
* Tracheoesophageal
* Bronchoesophageal
* Gastric, duodenal, jejunal, ileal, colonic or anastomotic -communicating to the skin (cutaneous)
* Esophogealgastric anastomosis
* Mediastinal anastomotic leak
* Fistula etiology may include:
* Secondary to previous malignancy with complete remission
* Secondary to radiotherapy as long as complete remission for 5 years has been achieved and documented
* Congenital with or without previous treatment
* Secondary to surgical interventions or endoscopic therapies such as dilation and esophageal manipulation
* Post prolonged tracheal intubation
* Secondary to inflammatory bowel disease
* Secondary to foreign body ingestion
* Secondary to thoracic trauma/crush injuries
* Secondary to caustic ingestion
* Secondary to pneumonectomy or mechanical ventilation
* Esophagomalacia
* The ability of subjects to give appropriate consent or have an appropriate representative available to do so
* The ability of subjects to return for follow up endoscopic assessment as established.

Exclusion Criteria

* Exposure to any investigational drug or procedure within 3 months prior to study entry.
* Patients with allergy to fibrin glue (TISSEEL) or anesthetics
* Patients with active/ongoing malignancy such as esophageal, lung, tracheal, thyroid, oropharyngeal or gastric cancer
* Patients on active regimen of chemotherapy
* Patients receiving radiation
* Diabetics with poor glucose metabolic control exhibited by an HbA1c > 9
* If there is evidence, in endoscopy, of dysplastic-appearing mucosa such as Barrett's dysplasia near the fistula or sinus tracts, this will be excluded. Patients that require surgical intervention at the fistula or sinus tract area for any reason
* BMI of <16 (may difficult lipoaspiration procedure)
* Women who are pregnant or nursing or women of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Clinical signs of respiratory tract or pleuro-pulmonary infections
* Prolonged (> 6 months) use of steroids
* Patients with fistulae or sinus tracts >15mm
* Drug or alcohol dependence
* Active infectious disease positive for HIV, HTLV, HBV, HCV, CMV (IgM > IgG) and/or syphilis
* End of life

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of Adverse Events from a single dose of autologous stromal vascular fraction (SVF) applied endoscopically into aerodigestive fistulae or enterocutaneous fistula [Safety and Tolerability]. | 5 Years
  Documentation of signs of adverse reactions from intravascular application of TISEEL, including: intravascular coagulation, thromboembolic events and acute hypersensitivity reactions. Documentation of signs of increased fistula size and/or aggravation of symptoms associated with fistulous tract, including: paroxysmal cough, dysphagia, wheezing, abdominal distention, chest pain, dyspnea, pneumonia.
Assessment of Adverse Events from liposuction procedure [Safety and Tolerability]. | 5 Years
  Signs of adverse reactions to the lipoaspiration procedure, including: allergic reaction to Hunstad solution, infection at the puncture wound site or risk of bleeding at the puncture wound site.

SECONDARY OUTCOMES:
Assessment of efficacy of Stromal Vascular Fraction's (SVF)'s ability to improve the success of surgical repair by fistulous tract reduction and/or closure. | 16 weeks
  Measurement and photography of the fistula in endoscopic/bronchoscopic evaluation.
Assessment of efficacy of Stromal Vascular Fraction's (SVF)'s ability to improve the success of surgical repair in reducing cardinal symptoms. | 5 Years
  Documentation of reduction of cardinal symptoms by history and physical examination.
Assessment of efficacy of Stromal Vascular Fraction's (SVF)'s ability to prevent recurrence of aerodigestive fistulae or enterocutaneous fistulae. | 5 Years
  Documentation of fistula recurrence by long term follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Bhaumik Brahmbhatt, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT03792360/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT03792360/ICF_001.pdf